CLINICAL TRIAL: NCT04580979
Title: A Natural History Study of Neurodegeneration and Optic Atrophy Caused by Ferredoxin Reductase Mutations in Pediatric and Adult Patients
Brief Title: Natural History Study of FDXR Mutation-related Mitochondriopathy
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: The Callum McKeefery and Nikki Albano McKeefery Pediatric Division of Genetics Fund (Unknown)
Responsible Party: Principal Investigator, Taosheng Huang, Principal Investigator, State University of New York at Buffalo
Other Study IDs: STUDY00004513-FDXR
Record Dates: First submitted 2020-10-02; First posted 2020-10-09 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Neurodegenerative Disease, Hereditary; Mitochondrial Diseases; Optic Atrophy
Keywords: Neurodegeneration; Mitochondrial disease; Optic atrophy; Ferredoxin reductase; Iron-sulfur cluster biogenesis; Iron overload; Iron homeostasis
MeSH Terms: conditions — Heredodegenerative Disorders, Nervous System; Mitochondrial Diseases; Optic Atrophy; Nerve Degeneration; Iron Overload

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — The medical records will be retained for all patients. For select patients, blood, DNA, skin punch biopsies will also be obtained for the purpose of genetic and biochemical analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with ferredoxin reductase deficiency: Male and female patients from age 2 to age 65 with clinically confirmed FDXR mutations. Both living and deceased patients will be included, if eligible. For deceased patients, the patient's medical history records will be reviewed, and an interview of the parent(s) or caregiver(s) will be performed.
  Interventions: Genetic: Mutation analysis

INTERVENTIONS:
Genetic: Mutation analysis — The investigators will sequence DNA samples from the patients or their families.

SUMMARY:
The purpose of the study is to systematically characterize the clinical course of the progressive neuropathy and optic atrophy observe in pediatric and adult patients with biallelic mutations in the ferredoxin reductase gene.

DETAILED DESCRIPTION:
The mitochondrial membrane-associated ferredoxin reductase (FDXR) is a flavoprotein that initiates the mitochondrial electron transport chain by transferring electrons from NADPH to the mitochondrial cytochrome P450 system via the ferredoxins FDX1 or FDX2. In addition to essential roles in Fe-S cluster biogenesis, this pathway is also central to the biosynthesis of steroid hormones. Previously, Dr. Taosheng Huang's research group has identified mutations in the FDXR gene in many individuals who share clinical presentations consistent with a mitochondrial disorder-including ataxia, hypotonia and optic atrophy-and obtained a naturally-occurring Fdxr mutant mouse model from Jackson Lab that corroborated these results (PMID: 29040572 and PMID: 30250212). In particular, FDXR enzyme activity, mitochondrial complex activities and ATP production were all significantly reduced in their patient samples. Their studies further indicated that Fdxr mutation leads to neurodegeneration that is associated with both inflammation as well as the abnormal accumulation of iron in the mitochondria, likely as a result of disrupted Fe-S cluster synthesis. More recently, his group has used the CRISPR-Cas9 system to generate a mouse line with a p.R389W amino acid change, which more precisely matches the most common human variant observed in their patients and shows a much more severe phenotype than their previous, naturally occurring Fdxr mouse model. They have also show that AAV-based gene therapy can significantly improve the condition of Fdxr mutant mice (DOI:https://doi.org/10.1016/j.omtm.2020.05.021), providing valuable preclinical data that may open the door for adapting such gene therapy treatments for use in human clinical trials. Given the recent regulatory approval granted to gene therapy treatments for LCA2, SMA1, and β-thalassemia, there is strong possibility that such an approach will ultimately produce a viable clinical treatment for FDXR patients as well.

FDXR is required for Iron-sulfur (Fe-S) clusters synthesis which is essential for multiple important biological processes, including electron transfer, cofactor synthesis, and gene regulation. Fe-S cluster biosynthesis is a tightly regulated process that requires coordinated delivery of both iron and sulfur and is a cofactor of many proteins. A variety of human disorders have been associated with impaired Fe-S cluster synthesis, including neurodegenerative disorders (e.g. Friedreich's ataxia) and myopathy with lactic acidosis. Iron homeostasis, which requires precise synthesis and localization of Fe-S clusters in mitochondria, is critical to ensure that there is sufficient iron for cellular functions, without reaching toxic levels of iron. Excessive levels of iron favor the formation of excess oxygen free radicals and consequent mitochondrial dysfunction.

The Rare Disease Act and Rare Disease Orphan Product Development Act highlight the importance of rare disease research and the obstacles to developing effective treatments for these diseases. However, the study of rare diseases may open a window to studying other human conditions. For example, Iron-sulfur biosynthesis abnormalities have been observed in more common human diseases such as Friedreich's ataxia. This relationship highlights the importance of human disease research by multiple approaches to understand biological mechanisms and for general application to human health. For these reasons, a better understanding of the pathogenesis of FDXR deficiency may help facilitate our knowledge of disease biology, neurodevelopment, brain function, and other organ abnormalities. Thus, in order to better understand the function of FDXR and to help lay the groundwork for eventual clinical trials of gene therapy or drug-based treatments for FDXR-related disease, the investigators propose this natural history study of both pediatric as well as adult patients with biallelic mutations in the ferredoxin reductase gene.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are clinically diagnosed with biallelic mutations in the ferredoxin reductase gene
* Male and female patients from 2 to 65 years of age
* Patients who have consented to the study
* In the case of a deceased patient whose parent(s) and/or legal guardian(s) have provided informed consent for study participation, the investigators will review the patient's medical records to determine study eligibility.

Exclusion Criteria:

* Significant postnatal complications or congenital anomalies that are not known to be associated with ferredoxin reductase deficiency
* Patient has received any experimental treatment for ferredoxin reductase deficiency within the 6 months prior to enrollment, or is expected to receive any such therapy during the study period

Ages: 0 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
Custom Medical History Questionnaire for Patients with FDXR Mutation-related Mitochondriopathy | 3 years
  In addition to a standard medical history, patients or their legal guardians will be asked to complete a custom medical history questionnaire tailored toward conditions commonly observed in patients with biallelic FDXR mutations. The items that will be asked about in this questionnaire are as follows:
  1. Known mutations in FDXR
  2. Any family history of illness
  3. Complications of pregnancy
  4. Premature birth
  5. Complications with birth
  6. Developmental delay
  7. Developmental regression
  8. Abnormal size of brain
  9. Movement disorders (ataxia, dystonia, etc.)
  10. Seizures
  11. Optic atrophy in eye exam
  12. Vision loss
  13. Other vision problems (color, eye movement)
  14. Hypotonia (muscle weakness or lack of tone)
  15. Electromyogram (EMG)
  16. Muscle biopsy
  17. Spasticity (muscle stiffness or tightness)
  18. Brain MRI performed?
  19. Electroencephalogram (EEG)
Retrospective examination of the medical records of patients with FDXR Mutation-related Mitochondriopathy | 3 years
  With the informed consent of the patients or their parent(s) and/or legal guardian(s), the investigators will perform a retrospective examination of the medical records of both living and deceased patients with confirmed biallelic FDXR mutations.
Eye assessments to evaluate ocular health | 3 years
  Visual acuity examination will be performed to determine the patient's clarity or sharpness of vision.
Growth and development (height) | 3 years
  World Health Organization (WHO) growth charts will be used to document height in centimeters (cm) for patients ranging from ages 5 to 19 years old. Routine methods will be used to document height for all other age groups.
Growth and development (weight) | 3 years
  World Health Organization (WHO) growth charts will be used to document weight in kilograms (kg) for pediatric patients age 5 to 10 years old. Routine methods will be used to document weight for all other age groups.
Growth and development (BMI) | 3 years
  World Health Organization (WHO) growth charts will be used to document Body Mass Index (BMI) in kilograms per meter square for patients age 5 to 19 years old. Routine methods will be used to document BMI for all other age groups.
ACTH stimulation testing for adrenal insufficiency | 3 years
  FDXR is known to support the catalytic activities of steroidogenic enzymes involved in aldosterone and cortisol synthesis. However, this deficiency may be partial and therefore only manifest in situations with severe stress, putting these persons at risk for an adrenal crisis. Therefore, we will also be testing patients with pathogenic FDXR variants for their risk of an adrenal crisis using the well-established ACTH stimulation test, assessing their stress-response ability to produce aldosterone and cortisol by comprehensive steroid profiling from blood.

CONTACTS AND LOCATIONS:
Overall Officials: Taosheng Huang, Principal Investigator — State University of New York at Buffalo
Locations (1):
- UBMD Pediatrics, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slone J, Peng Y, Chamberlin A, Harris B, Kaylor J, McDonald MT, Lemmon M, El-Dairi MA, Tchapyjnikov D, Gonzalez-Krellwitz LA, Sellars EA, McConkie-Rosell A, Reinholdt LG, Huang T. Biallelic mutations in FDXR cause neurodegeneration associated with inflammation. J Hum Genet. 2018 Dec;63(12):1211-1222. doi: 10.1038/s10038-018-0515-y. Epub 2018 Sep 25. PMID 30250212
- [Background] Slone JD, Yang L, Peng Y, Queme LF, Harris B, Rizzo SJS, Green T, Ryan JL, Jankowski MP, Reinholdt LG, Huang T. Integrated analysis of the molecular pathogenesis of FDXR-associated disease. Cell Death Dis. 2020 Jun 4;11(6):423. doi: 10.1038/s41419-020-2637-3. PMID 32499495
- [Background] Peng Y, Shinde DN, Valencia CA, Mo JS, Rosenfeld J, Truitt Cho M, Chamberlin A, Li Z, Liu J, Gui B, Brockhage R, Basinger A, Alvarez-Leon B, Heydemann P, Magoulas PL, Lewis AM, Scaglia F, Gril S, Chong SC, Bower M, Monaghan KG, Willaert R, Plona MR, Dineen R, Milan F, Hoganson G, Powis Z, Helbig KL, Keller-Ramey J, Harris B, Anderson LC, Green T, Sukoff Rizzo SJ, Kaylor J, Chen J, Guan MX, Sellars E, Sparagana SP, Gibson JB, Reinholdt LG, Tang S, Huang T. Biallelic mutations in the ferredoxin reductase gene cause novel mitochondriopathy with optic atrophy. Hum Mol Genet. 2017 Dec 15;26(24):4937-4950. doi: 10.1093/hmg/ddx377. PMID 29040572
- [Background] Yang L, Slone J, Zou W, Queme LF, Jankowski MP, Yin F, Huang T. Systemic Delivery of AAV-Fdxr Mitigates the Phenotypes of Mitochondrial Disorders in Fdxr Mutant Mice. Mol Ther Methods Clin Dev. 2020 May 22;18:84-97. doi: 10.1016/j.omtm.2020.05.021. eCollection 2020 Sep 11. PMID 32995353
- [Background] Campbell T, Slone J, Metzger H, Liu W, Sacharow S, Yang A, Moosajee M, La Morgia C, Carelli V, Palombo F, Lines MA, Innes AM, Levy RJ, Neilson D, Longo N, Huang T. Clinical study of ferredoxin-reductase-related mitochondriopathy: Genotype-phenotype correlation and proposal of ancestry-based carrier screening in the Mexican population. Genet Med Open. 2023 Nov 11;2:100841. doi: 10.1016/j.gimo.2023.100841. eCollection 2024. PMID 39669623